CLINICAL TRIAL: NCT01031173
Title: An Open-label Treatment Protocol to Evaluate the Safety of Replagal Treatment in Patients With Fabry Disease.
Brief Title: Treatment Protocol of Replagal for Patients With Fabry Disease
Status: No longer available | Type: Expanded Access
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Other Study IDs: HGT-REP-059; NCT00726089 (obsolete NCT alias)
Record Dates: First submitted 2009-12-08; First posted 2009-12-14 (Estimated); Last update posted 2021-05-24 (Actual); Status verified 2021-05

CONDITIONS: Fabry Disease
Keywords: α galactosidase A; glycosphingolipid storage disorder; agalsidase alfa; enzyme replacement therapy; Replagal; agalsidase beta; Fabrazyme
MeSH Terms: conditions — Fabry Disease | interventions — agalsidase alfa

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Biological: agalsidase alfa — 0.2 mg/kg body weight, administered by an intravenous infusion over 40 minutes, every other week.
  Other Names: Replagal

SUMMARY:
The study will evaluate the safety and efficacy of Replagal® (agalsidase alfa) at a dose of 0.2 mg/kg infused intravenously (IV) over 40 minutes, every other week. The study will monitor the course of disease in males and females with Fabry disease who are naive to treatment or were previously treated with agalsidase beta (Fabrazyme®).

DETAILED DESCRIPTION:
This study will evaluate the safety and efficacy of Replagal in patients with Fabry disease who are either naive to treatment, who were previously treated with agalsidase beta, or who had previously received Replagal.

Patients diagnosed with Fabry disease who have not previously received treatment, who have received agalsidase beta, or who had previously received Replagal will be eligible to enroll in the study and will receive Replagal at a dose of 0.2 mg/kg body weight administered by an IV infusion over 40 minutes every other week.

This study will be conducted in the United States.

Study visits will occur in 3 phases:

* Screening/Baseline Phase: A Screening/Baseline period (Day -30 to Day -1) to determine eligibility and obtain baseline measurements. Patients who have previously received agalsidase beta will be tested for the presence of anti-agalsidase beta antibodies.
* Treatment Phase: A 12-month treatment phase during which all patients will receive Replagal administered IV every other week. Clinical assessments will occur at Months 1, 3, 6, 9, and 12. The study may be extended to continue giving patients access to treatment.
* End-of-Study Phase: An end-of-study contact either as an office visit or follow-up telephone call will occur one month after the last infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of Fabry disease.
2. Patient is willing and able to provide written informed consent, and assent if applicable.
3. Females of childbearing potential must agree to use a method of birth control throughout the study and for at least 30 days after the final infusion. The method of contraception must be considered adequate and appropriate in the opinion of the investigator.

Exclusion Criteria:

1. Hypersensitivity to Replagal, the active substance, or any of the excipients.
2. The patient is pregnant or breast feeding.
3. Concomitant use of agalsidase beta (Fabrazyme).
4. Has received treatment with any investigation drug or device within the 30 days prior to study entry.
5. Otherwise unsuitable for the study, in the opinion of the Investigator.

Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (25):
- United States (25):
  - AKDHC Tucson Campbell, Tucson, Arizona
  - University of California San Diego Medical Center, La Jolla, California
  - Kaiser Medical Group Southern CA, Regional Metabolic Services, Los Angeles, California
  - Children's Hospital & Research Center Oakland, Oakland, California
  - UC Davis Children's Hospital, Sacramento, California
  - Central Coast Nephrology, Salinas, California
  - Denver Nephrologists, PC, Denver, Colorado
  - University Research Foundation for Lysosomal Storage Disorders, Coral Springs, Florida
  - Stuart Oncology Associates, Stuart, Florida
  - Emory University School of Medicine, Decatur, Georgia
  - Emory University, Decatur, Georgia
  - University of Iowa Health Center, Iowa City, Iowa
  - Baystate Medical Center, Springfield, Massachusetts
  - Infusion Associates, Grand Rapids, Michigan
  - University of Missouri Healthcare, Columbia, Missouri
  - St. Joseph's Regional Medical Center, Paterson, New Jersey
  - North Shore Hematology/Oncology, Manhasset, New York
  - New York University School of Medicine, New York, New York
  - Fullerton Genetics Center-Mission, St. Joseph's Hospital, Asheville, North Carolina
  - The Toledo Hospital, Toledo, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Baylor University Medical Center, Dallas, Texas
  - Tidewater Kidney Specialists, Chesapeake, Virginia
  - Carilion New River Valley Medical Center, Christiansburg, Virginia
  - O & O Alpan LLC, Springfield, Virginia